CLINICAL TRIAL: NCT05609422
Title: Effect of Scooter Board Activities on Trunk Postural Control and Gait in Children With Diplegic Cerebral Palsy
Brief Title: Scooter Board Activities in Diplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Omnya Samy Abdallah Ghoneim, Lecturer, Department of Physical Therapy for Pediatrics and Pediatric Surgery, Faculty of Physical Therapy, Badr University in Cairo, Egypt., Badr University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Omnya 2
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Diplegia
Keywords: diplegia; cerebral palsy; core stability; trunk control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The selected subjects will be divided into two groups of equal numbers (control and study).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Received the designed physical therapy program.
  Interventions: Other: Physical therapy program
- study group (Experimental): Received a designed physical therapy program in addition to scooter bord activities.
  Interventions: Other: Physical therapy program; Other: scooter board activities

INTERVENTIONS:
Other: Physical therapy program — * Stretching exercises
  * Strength Training Kneeling exercises
  * Standing exercises
  * Gait Training
Other: scooter board activities — 1. Scooter board bear walk.
  2. Scooter board crab walk.
  3. Sitting on scooter board, use it to move forward and backward, move the pool rings from one end to another.
  4. Cross sitting on scooter board, pulls along the rope using his/her hands
  5. Sit with knees pulled into the chest (like a bug pose) and move around with arms only.
  6. Prone over scooter board, pulling rope to move forward. Pull self along an anchored rope to retrieve items
  7. Scooter rolls outs. Place knees on floor and hands holding the edge of the front scooter board. Push board out a few inches then pull back, the further you roll, the harder it gets.
  8. Kneeling, Push self forward and backward with the use of a therapy ball (lots of Motor Planning).
  9. Supine flexion on scooter board, Clip clothespins to a rope hanging above.
  Arms: study group

SUMMARY:
Children with CP may have muscle weakness, changes in mobility, posture, muscle tone, motor coordination and deficits in postural control. These changes, individually or collectively, affect psychomotor function. As a result, activities that are performed quickly and readily by healthy children may be difficult and time-consuming for children with CP.

DETAILED DESCRIPTION:
Similar vestibular stimulation can be provided with ascooter-board which requires more active participation on the part of the child. A scooter-board is simply a wooden board mounted on four castors so that it can roll freely and spin in any direction, it should be big enough to support the middle part of the body while the head, upper chest and legs hang off the ends.

ELIGIBILITY:
Inclusion Criteria:

1. CP with a diplegia
2. Age 7 to 11 years
3. Grade 1and 2 according to the Modified Ashworth scale (RW and Smith, 1987).
4. They could walk with limitation or holding on according to GMFCS (level I&II &III) (Palisano et al., 1997).
5. They were able to understand and follow verbal instructions

Exclusion Criteria:

1. Children with any surgical interference in the upper limb.
2. intellectual disability such that simple tasks could not be understood or executed.
3. Children with any visual or auditory problems.
4. Children with any surgical interference in the lower limb.
5. Children with any structural deformities in joints and bones of lower limbs.
6. Children who suffer from other diseases or associated disorders that interfered with physical activity.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
Trunk control measurement scale (TCMS) | 3 months
  TCMS measures trunk control in two basic components:
  static and dynamic sitting balance. Balance is assessed during flexion, extension, lateral flexion, and rotation movements as selective movements of dynamic sitting. Total score ranges between 0 and 58, and higher scores indicate better control
2D video-based gait assessment system | 3 months
  2D video-based gait assessment system to measure lateral trunk sway at SLS from frontal view

CONTACTS AND LOCATIONS:
Overall Officials: Omnya samy, PHD, Principal Investigator — lecturer
Locations (1):
- Badr University, Badr, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Private data for this research